CLINICAL TRIAL: NCT00940212
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Oral AZD2423 After Single Ascending Doses in Healthy Male and Female Volunteers Without Childbearing Potential
Brief Title: Study to Investigate Safety, Tolerability and Pharmacokinetics of AZD2423 in Healthy Volunteers
Acronym: SAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Anders Neijber, Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D2600C00001; EudraCT 2009-010364-42
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Healthy Volunteers
Keywords: Safety; tolerability; healthy; pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): AZD2423
  Interventions: Drug: AZD2423
- B (Experimental): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2423 — oral, single administration
  Arms: A
Drug: Placebo — oral administration and single dose
  Arms: B

SUMMARY:
The primary aim of this study is to investigate the safety and tolerability of AZD2423 single doses in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Have a body mass index (BMI) between ≥18 and ≤30 kg/m2, as calculated by the investigator, and weigh at least 50 kg and no more than 100 kg
* Healthy male and non-fertile female volunteers with suitable veins for cannulation or repeated venipuncture

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study,or influence the results or the subject's ability to participate in the study
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Any clinically significant illness/infection or medical/surgical procedure or trauma,as judged by the Principal Investigator, within 3 months of the first administration of investigational product

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of AZD2423 following administration of single ascending doses and if possible to estimate the maximum tolerated dose (MTD), if within the predefined exposure limits. | 3 day residential period plus 7-10 days follow up

SECONDARY OUTCOMES:
To characterise the pharmacokinetics of AZD2423 and provisionally assess the dose proportionality of the pharmacokinetics following administration of single ascending doses ofAZD2423. | 3 day residential period plus 7-10 days follow up

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, MD, Principal Investigator — PAREXEL Early Phase Clinical Uniit, Berlin Germany; Anders Neijber, Study Director — AstraZeneca R&D Södertälje
Locations (1):
- Research Site, Berlin, Germany